CLINICAL TRIAL: NCT04219969
Title: Ideal Imaging Time Point Assessment for Spinal Cord Lesions of Unknown Etiology With FDG PET-MRI
Brief Title: FDG PET-MRI for the Diagnosis of Spinal Cord Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018-0144; NCI-2019-08224 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0144 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-12-30; First posted 2020-01-07 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Spinal Cord Neoplasm
MeSH Terms: conditions — Spinal Cord Neoplasms | interventions — Fluorodeoxyglucose F18; Magnetic Resonance Imaging; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic (18F-FDG PET-MRI) (Experimental): Patients receive fludeoxyglucose F-18 IV over 1 minutes and then undergo PET-MRI over 15-60 minutes at 60, 300, and 480 minutes after fludeoxyglucose F-18 injection in the absence of unacceptable toxicity.
  Interventions: Drug: Fludeoxyglucose F-18; Device: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography

INTERVENTIONS:
Drug: Fludeoxyglucose F-18 — Given IV
  Other Names: 18FDG; FDG; Fludeoxyglucose (18F); fludeoxyglucose F 18; Fludeoxyglucose F18; Fluorine-18 2-Fluoro-2-deoxy-D-Glucose; Fluorodeoxyglucose F18
Device: Magnetic Resonance Imaging — Undergo PET-MRI
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; nuclear magnetic resonance imaging
Procedure: Positron Emission Tomography — Undergo PET-MRI
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging

SUMMARY:
To compare the results and understand the possible benefits from FDG-PET/MRI during different scanning time points after FDG, a type of contrast drug, is given.

DETAILED DESCRIPTION:
Primary Objectives:

--To identify the optimal imaging time point using F18-FDG positron emission tomography (PET) that gives the best lesion conspicuity as defined by the best lesion to background (L/B) ratio when evaluating spinal cord lesions of unknown etiology.

Exploratory Objectives:

* To identify malignancy specific factors in F18-FDG metabolism derived from metrics such as maximum standard uptake value (SUVmax), mean standard uptake value (SUVmean), total lesion glycolysis (TLG), metabolic tumor volume (MTV) and L/B ratio.
* To identify patterns of metabolism derived from metrics such as SUVmax, SUVmean, TLG, MTV, L/B ratio and magnetic resonance imaging metrics such as regional perfusion abnormalities, apparent diffusion coefficient values and mean diffusivity measures.

OUTLINE:

Patients receive fludeoxyglucose F-18 intravenously (IV) over 1 minutes and then undergo PET-magnetic resonance imaging (MRI) over 15-60 minutes at 60, 300, and 480 minutes after fludeoxyglucose F-18 injection in the absence of unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with untreated intramedullary cord lesion(s)
* Ability to undergo FDG PET MR examination

Exclusion Criteria:

* No prior surgery or biopsy of the spinal cord
* No metal implanted in area of interest
* Spine radiation therapy
* Known allergy to FDG or gadolinium based contrast agents
* Blood glucose (> 200 mg/dl)
* Pregnant women are excluded
* Children of less than 18 years of age
* Need for conscious sedation or anesthesia in order to tolerate study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-09-21 (Actual); Primary Completion 2024-05-07 (Actual); Study Completion 2024-05-07 (Actual)

PRIMARY OUTCOMES:
Standard uptake value (SUV) max | Up to 8 hours
  Identifying the specific malignancy
Lesion to background (L/B) ratio | Up to 8 hours
  L is the lesion metric (mean, max, etc.) and B is the corresponding background metric. These values will be plotted versus time and the delayed time point corresponding to the highest value for each metric recorded. Differences in L/B ratio will be tested via paired t-test.
Optimal imaging time point | Up to 8 hours
  Defined as the time point by which there is the largest average SUVmax L/B ratio and significantly different from baseline at the 0.025 significance level.

CONTACTS AND LOCATIONS:
Overall Officials: Maria K Gule-Monroe, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org